CLINICAL TRIAL: NCT06928805
Title: Determination of the Effects of Two Different Breathing Techniques and Forward-Leaning Position on Physiological Parameters in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: The Effects of Two Different Breathing Techniques and Forward-Leaning Position on Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SaglikBilimleriU Semra Aciksoz
Record Dates: First submitted 2025-03-28; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease, COPD
Keywords: Chronic Obstructive Pulmonary Disease; Breathing Techniques; Forward-Leaning Position; Physiological Parameters
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pursed-lip breathing exercise (Experimental)
  Interventions: Other: Pursed-lip breathing exercise
- Balloon inflation exercise (Experimental)
  Interventions: Other: Balloon inflation exercise
- Standard treatment (Experimental)
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: Balloon inflation exercise — Balloon inflation exercise was applied in addition to the forward-leaning position.
  Arms: Balloon inflation exercise
Other: Pursed-lip breathing exercise — The pursed-lip breathing exercise was applied in addition to the forward-leaning position.
  Arms: Pursed-lip breathing exercise
Other: Control (Standard treatment) — Standard practice is implemented in the institution where the study is conducted.
  Arms: Standard treatment

SUMMARY:
This study aims to determine the effects of balloon inflation and pursed-lip breathing exercises, in addition to the forward-leaning position, on physiological parameters in individuals with Chronic Obstructive Pulmonary Disease (COPD).

The hypotheses of the study are as follows:

H1_1: The forward-leaning position and balloon inflation breathing exercise have a positive effect on physiological parameters in patients with Chronic Obstructive Pulmonary Disease (COPD).

H1_2: The forward-leaning position and pursed-lip breathing exercise have a positive effect on physiological parameters in patients with COPD.

H1_3: There is a significant difference in physiological parameters between the balloon inflation and pursed-lip breathing exercise groups and the control group.

Within this scope, the study will be conducted with three groups:

Intervention Group 1: Balloon inflation exercise applied in addition to the forward-leaning position.

Intervention Group 2: Pursed-lip breathing exercise applied in addition to the forward-leaning position.

Control Group: Standard practice implemented in the institution where the study is conducted.

Participants:

* A home exercise program will be designed for both intervention groups, allowing them to perform the exercises independently each day.
* The exercises will start with three sessions per day and will be increased by one session each week, continuing for a total of four weeks.
* Participants will visit the outpatient clinic in the 4th week for assessments and tests.
* Patients will be contacted weekly by the researcher via phone to ensure adherence to the program.

DETAILED DESCRIPTION:
The exercise program will be determined in collaboration with a respiratory physiotherapist and implemented by the researcher. Accordingly, patients with stage II-III COPD (as determined by a physician) who visit the pulmonology outpatient clinic of the relevant hospital and meet the inclusion criteria will be given brief information about respiratory exercises, their benefits, and duration. They will then be instructed on how to perform the exercises through verbal commands for approximately 30 minutes. At the end of the session, the exercise guidelines will be practiced under the supervision of the researcher.

Before starting, the patient will be seated in a chair and allowed to rest for about 15 minutes. The patient will be informed about how to perform the walking test, the expected walking pace, and that they can stop and rest if they feel fatigued. Then, the patient will be asked to walk at a brisk pace for six minutes under the supervision of the researcher. During the walk, the researcher will continuously monitor the patient's oxygen saturation using a handheld pulse oximeter. If the patient exhibits signs of excessive sweating, pallor, or a significant drop in oxygen levels, the test will be terminated early.

Before and after the test, blood pressure, pulse rate, respiratory rate, oxygen saturation [SpO2], and dyspnea score using the Modified Borg Scale will be assessed, and the distance the patient walks in six minutes will be recorded. The six-minute walk test will be repeated at the end of the study. Subsequently, the patient will undergo a pulmonary function test, and the values for FVC, FEV1, FEV1/FVC ratio, and peak expiratory flow will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have no communication and cooperation problems,
* Can speak and understand Turkish,
* Have a baseline saturation of >90%,
* Have been diagnosed with Stage II and Stage III COPD,
* Have not had any infection or COPD exacerbation for at least 3 months,
* Have not participated in a pulmonary rehabilitation program in the last 3 months,
* Can walk without assistance,
* Do not have serious and/or unstable heart disease, neuromuscular disease, orthopedic disease or mental illness that may impair their physical activities of daily living,
* Willing to participate in the study will be included.

Exclusion Criteria:

* Patients who have been hospitalized since the start of the study,
* Those receiving continuous oxygen therapy,
* Those who have cooperation problems,
* Those who cannot adapt to exercise,
* Those who have 2-3 or more acute attacks per year,
* Those with a history of pulmonary hypertension, malignancy, pulmonary thromboembolism, obstructive sleep apnea, unstable angina or myocardial infarction,
* Patients with a pulse rate over 120/minute will be excluded from the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
blood pressure | 4 weeks later
pulse | 4 weeks later
respiratory rate | 4 weeks later
saturation | 4 weeks later

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | 4 weeks later
Forced Expiratory Volume in One Second (FEV1) | 4 weeks later
FEV1/FVC ratio | 4 weeks later
Peak Expiratory Flow (PEF) | 4 weeks later
Modified Borg Dyspnea Scale (MBS) | 4 weeks later
  MBS determines the severity of dyspnea at rest and during exertion. It consists of 10 items that define the severity of dyspnea according to its degree. A score of 0 indicates no dyspnea, and a score of 10 indicates very severe dyspnea.
6 Minute Walking Test (6MWT) | 4 weeks later
  The test evaluates functional exercise capacity by measuring the distance in meters that the patient will cover in 6 minutes by walking as fast as possible but without running in a 30-meter uninterrupted corridor.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Aciksoz, RN, Assistant Professor, PhD, Principal Investigator — University of Health Sciences Turkey, Hamidiye Faculty ofNursing
Locations (1):
- University of Health Sciences Turkey, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided